CLINICAL TRIAL: NCT06654089
Title: A Real-World Evidence Study Evaluating Quality of Life Parameters Following Use of Emergen-C
Brief Title: A Study Evaluating Quality of Life Parameters Following Use of Emergen-C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 300217
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emergen-C Core Super Orange Powder (Test Product) (Experimental): Participants will be instructed to take the study product as per label instructions. Participants will consume one sachet of Emergen-C Core Super Orange Powder stirred in 4-6 ounces of water, orally, once daily for up to 12 weeks.
  Interventions: Dietary Supplement: Emergen-C Core Super Orange Powder
- Placebo (Reference Product) (Placebo Comparator): Participants will be instructed to take the study product as per label instructions. Participants will consume one sachet of placebo stirred in 4-6 ounces of water, orally, once daily for up to 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Emergen-C Core Super Orange Powder — A dietary supplement powder containing vitamin C, zinc, vitamin B6, vitamin B12, folate, and manganese.
  Arms: Emergen-C Core Super Orange Powder (Test Product)
Dietary Supplement: Placebo — A study product identical to the test product without active ingredients.
  Arms: Placebo (Reference Product)

SUMMARY:
The purpose of this study is to determine how Emergen-C use can improve quality of life (QoL) in a real-world setting to help consumers and healthcare professionals understand the benefits of taking Emergen-C on a routine or daily basis.

DETAILED DESCRIPTION:
This will be a randomized, double-blinded, placebo-controlled clinical trial to evaluate the over-time effects of 12-weeks Emergen-C supplementation on QoL parameters in a real-world setting. This study will be entirely decentralized, and participants will not be required to physically attend any on-site visits. All study data will be collected remotely through a study platform using the participant's personal mobile device, tablet or computer. Sufficient participants will be screened to enroll approximately 300 eligible participants (approximately 150 participants per group) and approximately 240 participants are expected to complete the study (approximately 120 participants per group).

ELIGIBILITY:
Inclusion Criteria:

* Participant's provision of a signed and dated electronic informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Healthy adults, 18-64 years of age at the time of electronic consent (does not exclude any ethnicities, races, or gender identities).
* Participant is seeking to improve their energy/less fatigue levels.
* Participants whose baseline score is greater than or equal to (>=) 10 on the dimension of general fatigue of the MFI and a score >=3 for at least ten of the 20 questions of the MFI.
* Participants who are willing and able to comply with all study related activities as shown in the Schedule of Activities.
* Participants who reside in the United States (except for Hawaii and Alaska).
* Participants who own a mobile device, tablet or computer with access to stable internet connection and are willing to use their device to complete study surveys and assessments.

Exclusion Criteria:

* Participants who are either directly involved in the conduct of the study or a member of their immediate family; or a Haleon employee directly involved in the conduct of the study or a member of their immediate family.
* Participants who have participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days prior to study entry and/or during study participation.
* Participants who are pregnant, lactating, or plan to be pregnant or lactating during the course of the study (self-report).
* Participants with known or suspected intolerance or hypersensitivity to any study materials (or closely related compounds) or any of their stated ingredients.
* Participants who are hypertensive or salt-sensitive should be excluded from this study.
* Participants who report being a heavy drinker (defined as drinking 3 or more alcoholic beverages per day).
* Participants who are unable to read and understand English.
* Participants who report current and/or recent (up to 3 months ago) major illnesses and/ or major surgery.
* Participants who report a planned surgery during the study duration.
* Participants who report a diagnosis of heart failure, heart rhythm disturbances, severe liver disease, severe mental health diagnosis, or severe renal failure.
* Participants who report taking medications (in the previous 21 days) that have well established moderate or severe interaction with any of the study product ingredients: Anticoagulants, antihypertensives, anxiolytics, antidepressants, chemotherapy, immunotherapy, sedative hypnotics, medications that warn against grapefruit consumption, corticosteroids at doses greater than 5 milligrams (mg) per day, diabetic medications, oral anti-infectives (antibiotics, antifungals, antivirals) to treat an acute infection, antipsychotics, Monoamine Oxidase Inhibitors (MAOIs), or thyroid products.
* Participants who are currently taking a multivitamin or have taken a multivitamin in the past 30 days and are not willing to stop taking a multivitamin for the duration of the trial.
* Participants who are currently taking other Vitamin C or B supplements or have taken Vitamin C or B supplements in the past 30 days and are not willing to stop taking other Vitamin C or B supplements for the duration of the trial.
* Participants who are currently consuming energy drinks or energy shots or have consumed an energy drink or energy shot in the past 30 days and are not willing to stop consuming energy drinks and energy shots for the duration of the trial.
* A participant who has previously been enrolled in this study.
* A participant who, in the opinion of the investigator or delegate, should not participate in the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 299 (Actual)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Multidimensional Fatigue Inventory (MFI) General Fatigue Domain (Items 1,5,12,16) Score at Week 12 | Baseline and Week 12
  The MFI is a 20-item scale designed to evaluate five dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue. General fatigue domain has 4 items (Item 1: I feel fit; Item 5: I feel tired; Item 12: I am rested; Item 16: I tire easily). Participants will answer how they feel about each item, lately on a scale of 1 (yes, that is true) to 5 (no, that is not true). Positively phrased items will be reverse scored and negatively phrased items will be scored at face value. The total domain score will be calculated by summation of the scores of individual items and can range from 4 to 20 where lower scores indicate lower level of fatigue. Change from Baseline will be calculated by subtracting the Baseline score from score at Week 12. A negative change from Baseline will indicate improvement in fatigue.
Change from Baseline in MFI Physical Fatigue Domain (Items 2,8,14,20) Score at Week 12 | Baseline and Week 12
  The MFI is a 20-item scale designed to evaluate five dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue. Physical fatigue domain has 4 items (Item 2: Physically I feel only able to do a little; Item 8: Physically I can take on a lot; Item 14: Physically I feel I am in a bad condition; Item 20: Physically I feel I am in an excellent condition). Participants will answer how they feel about each item, lately on a scale of 1 (yes, that is true) to 5 (no, that is not true). Positively phrased items will be reverse scored and negatively phrased items will be scored at face value. The total domain score will be calculated by summation of the scores of individual items and can range from 4 to 20 where lower scores indicate lower level of fatigue. Change from Baseline will be calculated by subtracting the Baseline score from score at Week 12. A negative change from Baseline will indicate improvement in fatigue.
Change from Baseline in MFI Reduced Activity Domain (Items 3,6,10,17) Score at Week 12 | Baseline and Week 12
  The MFI is a 20-item scale designed to evaluate five dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue. Reduced activity domain has 4 items (Item 3: I feel very active; Item 6: I think I do a lot in a day; Item 10: I think I do very little in a day; Item 17: I get little done). Participants will answer how they feel about each item, lately on a scale of 1 (yes, that is true) to 5 (no, that is not true). Positively phrased items will be reverse scored and negatively phrased items will be scored at face value. The total domain score will be calculated by summation of the scores of individual items and can range from 4 to 20 where lower scores indicate lower level of fatigue. Change from Baseline will be calculated by subtracting the Baseline score from score at Week 12. A negative change from Baseline will indicate improvement in fatigue.
Change from Baseline in MFI Reduced Motivation Domain (Items 4,9,15,18) Score at Week 12 | Baseline and Week 12
  The MFI is a 20-item scale designed to evaluate five dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue. Reduced motivation domain has 4 items (Item 4: I feel like doing all sorts of nice things; Item 9: I dread having to do things; Item 15: I have a lot of plans; Item 18: I don't feel like doing anything). Participants will answer how they feel about each item, lately on a scale of 1 (yes, that is true) to 5 (no, that is not true). Positively phrased items will be reverse scored and negatively phrased items will be scored at face value. The total domain score will be calculated by summation of the scores of individual items and can range from 4 to 20 where lower scores indicate lower level of fatigue. Change from Baseline will be calculated by subtracting the Baseline score from score at Week 12. A negative change from Baseline will indicate improvement in fatigue.
Change from Baseline in MFI Mental Fatigue Domain (Items 7,11,13,19) Score at Week 12 | Baseline and Week 12
  The MFI is a 20-item scale designed to evaluate five dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue. Mental fatigue domain has 4 items (Item 7: When I am doing something, I can keep my thoughts on it; Item 11: I can concentrate well; Item 13: It takes a lot of effort to concentrate on things; Item 19: My thoughts easily wander). Participants will answer how they feel about each item, lately on a scale of 1 (yes, that is true) to 5 (no, that is not true). Positively phrased items will be reverse scored and negatively phrased items will be scored at face value. The total domain score will be calculated by summation of the scores of individual items and can range from 4 to 20 where lower scores indicate lower level of fatigue. Change from Baseline will be calculated by subtracting the Baseline score from score at Week 12. A negative change from Baseline will indicate improvement in fatigue.

SECONDARY OUTCOMES:
Change from Baseline in MFI General Fatigue Domain (Items 1,5,12,16) Score at Weeks 4 and 8 | Baseline, Week 4 and Week 8
  The MFI is a 20-item scale designed to evaluate five dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue. General fatigue domain has 4 items (Item 1: I feel fit; Item 5: I feel tired; Item 12: I am rested; Item 16: I tire easily). Participants will answer how they feel about each item, lately on a scale of 1 (yes, that is true) to 5 (no, that is not true). Positively phrased items will be reverse scored and negatively phrased items will be scored at face value. The total domain score will be calculated by summation of the scores of individual items and can range from 4 to 20 where lower scores indicate lower level of fatigue. Change from Baseline will be calculated by subtracting the Baseline score from post-Baseline score at indicated timepoints. A negative change from Baseline will indicate improvement in fatigue.
Change from Baseline in MFI Physical Fatigue Domain (Items 2,8,14,20) Score at Weeks 4 and 8 | Baseline, Week 4 and Week 8
  MFI is a 20-item scale designed to evaluate five dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue. Physical fatigue domain has 4 items (Item 2: Physically I feel only able to do a little; Item 8: Physically I can take on a lot; Item 14: Physically I feel I am in a bad condition; Item 20: Physically I feel I am in an excellent condition). Participants will answer how they feel about each item, lately on a scale of 1 (yes, that is true) to 5 (no, that is not true). Positively phrased items will be reverse scored and negatively phrased items will be scored at face value. Total domain score will be calculated by summation of the scores of individual items and can range from 4 to 20 where lower scores indicate lower level of fatigue. Change from Baseline will be calculated by subtracting the Baseline score from post-Baseline score at indicated timepoints. A negative change from Baseline will indicate improvement in fatigue.
Change from Baseline in MFI Reduced Activity Domain (Items 3,6,10,17) Score at Weeks 4 and 8 | Baseline, Week 4 and Week 8
  The MFI is a 20-item scale designed to evaluate five dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue. Reduced activity domain has 4 items (Item 3: I feel very active; Item 6: I think I do a lot in a day; Item 10: I think I do very little in a day; Item 17: I get little done). Participants will answer how they feel about each item, lately on a scale of 1 (yes, that is true) to 5 (no, that is not true). Positively phrased items will be reverse scored and negatively phrased items will be scored at face value. The total domain score will be calculated by summation of the scores of individual items and can range from 4 to 20 where lower scores indicate lower level of fatigue. Change from Baseline will be calculated by subtracting the Baseline score from post-Baseline score at indicated timepoints. A negative change from Baseline will indicate improvement in fatigue.
Change from Baseline in MFI Reduced Motivation Domain (Items 4,9,15,18) Score at Weeks 4 and 8 | Baseline, Week 4 and Week 8
  The MFI is a 20-item scale designed to evaluate five dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue. Reduced motivation domain has 4 items (Item 4: I feel like doing all sorts of nice things; Item 9: I dread having to do things; Item 15: I have a lot of plans; Item 18: I don't feel like doing anything). Participants will answer how they feel about each item, lately on a scale of 1 (yes, that is true) to 5 (no, that is not true). Positively phrased items will be reverse scored and negatively phrased items will be scored at face value. The total domain score will be calculated by summation of the scores of individual items and can range from 4 to 20 where lower scores indicate lower level of fatigue. Change from Baseline will be calculated by subtracting the Baseline score from post-Baseline score at indicated timepoints. A negative change from Baseline will indicate improvement in fatigue.
Change from Baseline in MFI Mental Fatigue Domain (Items 7,11,13,19) Score at Weeks 4 and 8 | Baseline, Week 4 and Week 8
  The MFI is a 20-item scale designed to evaluate five dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue. Mental fatigue domain has 4 items (Item 7: When I am doing something, I can keep my thoughts on it; Item 11: I can concentrate well; Item 13: It takes a lot of effort to concentrate on things; Item 19: My thoughts easily wander). Participants will answer how they feel about each item, lately on a scale of 1 (yes, that is true) to 5 (no, that is not true). Positively phrased items will be reverse scored and negatively phrased items will be scored at face value. The total domain score will be calculated by summation of the scores of individual items and can range from 4 to 20 where lower scores indicate lower level of fatigue. Change from Baseline will be calculated by subtracting the Baseline score from post-Baseline score at indicated timepoints. A negative change from Baseline will indicate improvement in fatigue.
Change from Baseline in Individual Items (Items 1 to 20) Score in the MFI at Weeks 4, 8 and 12 | Baseline, Weeks 4, 8 and 12
  The MFI is a 20-item scale designed to evaluate five dimensions of fatigue: general fatigue (Items 1, 5, 12, 16), physical fatigue (Items 2, 8, 14, 20), reduced motivation (Items 4, 9, 15, 18), reduced activity (Items 3, 6, 10, 17), and mental fatigue (Items 7, 11, 13, 19). Participants will answer how they feel about each item, lately on a scale of 1 (yes, that is true) to 5 (no, that is not true). Positively phrased items will be reverse scored and negatively phrased items will be scored at face value. Each individual item score can range from 1 to 5 where lower scores indicate lower level of fatigue. Change from Baseline will be calculated by subtracting the individual MFI item score at Baseline from post-Baseline score at indicated timepoints. A negative change from Baseline will indicate improvement in fatigue.
Change from Baseline in Additional QoL Parameter at Weeks 4, 8 and 12: Family Support | Baseline, Weeks 4, 8 and 12
  Participants will answer 2 QoL questions (I feel more energized to look after my family and/or loved ones; I feel more prepared for the future) indicating how they feel about each statement, lately on a scale of 1 (yes, that is true) to 5 (no, that is not true). Lower scores indicate better quality of life. Change from Baseline will be calculated by subtracting the individual question score at Baseline from post-Baseline score at indicated timepoints. A negative change from Baseline will indicate improvement in quality of life.
Change from Baseline in Additional QoL Parameter at Weeks 4, 8 and 12: Resilience | Baseline, Weeks 4, 8 and 12
  Participants will answer 2 QoL questions (I feel resilient so I can be at my best each day; I feel ready to cope with life's challenges) indicating how they feel about each statement, lately on a scale of 1 (yes, that is true) to 5 (no, that is not true). Lower scores indicate better quality of life. Change from Baseline will be calculated by subtracting the individual question score at Baseline from post-Baseline score at indicated timepoints. A negative change from Baseline will indicate improvement in quality of life.
Change from Baseline in Additional QoL Parameter at Weeks 4, 8 and 12: Ability to Relax and Unwind | Baseline, Weeks 4, 8 and 12
  Participants will answer 2 QoL questions (I feel relaxed; I feel able to unwind) indicating how they feel about each statement, lately on a scale of 1 (yes, that is true) to 5 (no, that is not true). Lower scores indicate better quality of life. Change from Baseline will be calculated by subtracting the individual question score at Baseline from post-Baseline score at indicated timepoints. A negative change from Baseline will indicate improvement in quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Lindus Health Limited, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.